CLINICAL TRIAL: NCT00383032
Title: Randomized Controlled Trial of Mifepristone Versus Laminaria for Cervical Ripening In Midtrimester Induction
Brief Title: Mifepristone Versus Laminaria for Cervical Ripening in Midtrimester Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPHS # 16429
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2007-12

CONDITIONS: Abortion, Induced
MeSH Terms: interventions — Mifepristone

INTERVENTIONS:
Drug: mifepristone

SUMMARY:
Data from other countries have suggested that oral mifepristone used as a cervical ripening agent may decrease induction to delivery time in midtrimester inductions. To our knowledge, there are no trials comparing mifepristone to laminaria in a standard clinical setting with standardized misoprostol induction protocol to examine the issue of induction to delivery time. We hypothesize that mifepristone will work at least as well as laminaria for midtrimester cervical ripening prior to induction of labor with misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with fetal anomalies, aneuploidy, or demise at 15-22 weeks gestation
* age greater than 16
* able to speak English

Exclusion Criteria:

* prior uterine scar or
* allergy or history of bad reaction to any of the study drugs or
* history of chronic adrenal failure or
* porphyria or
* concurrent long-term corticosteroid treatment

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72
Dates: Start 2004-01; Study Completion 2006-06

PRIMARY OUTCOMES:
induction to delivery time

SECONDARY OUTCOMES:
pain
delivery within 24 hours
need for post-partum D&C
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Karen George, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Prairie BA, Lauria MR, Kapp N, Mackenzie T, Baker ER, George KE. Mifepristone versus laminaria: a randomized controlled trial of cervical ripening in midtrimester termination. Contraception. 2007 Nov;76(5):383-8. doi: 10.1016/j.contraception.2007.07.008. Epub 2007 Oct 4. PMID 17963864